CLINICAL TRIAL: NCT04447963
Title: Evaluation of Safety and Efficacy of the BTL-785F Device for Non-invasive Reduction of Wrinkles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTL-785F_WRI
Record Dates: First submitted 2020-06-22; First posted 2020-06-25 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Wrinkle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Non-invasive treatment of wrinkles and rhytids (Experimental): The subjects will be enrolled and assigned into one experimental study arm. The subjects will be required to complete three (3) treatment visits and two follow-up visits.
  At the baseline visit health status will be assessed and, if needed, additional tests will be performed. Inclusion and exclusion criteria will be verified and informed consent will be signed.
  The treatment administration phase consists of three (3) treatment visits, delivered 1 week apart.
  At every treatment visit after the first, prior to the procedure, the participants will be assessed for adverse effects resulting from the previous treatment(s) with the BTL-785F device.
  Interventions: Device: Non-invasive treatment of facial wrinkles

INTERVENTIONS:
Device: Non-invasive treatment of facial wrinkles — Application of radiofrequency field which provides controlled heating to the skin.Therapeutic effect is observed when the tissue temperature reaches 40-45 degrees Celsius.

SUMMARY:
This study will evaluate the clinical safety and the performance of the BTL-785F system equipped with BTL-785-2 applicator for non-invasive treatment of facial wrinkles.

DETAILED DESCRIPTION:
This study will evaluate the clinical safety and the performance of the BTL-785F system equipped with BTL-785-2 applicator for non-invasive treatment of facial wrinkles. The study is a multicenter single-arm, open-label, interventional study. The subjects will be enrolled and assigned into one experimental study arm. The subjects will be required to complete three (3) treatment visits and two follow-up visits. At every treatment visit after the first, prior to the procedure, the participants will be assessed for adverse effects resulting from the previous treatment(s) with the BTL-785F device.

Safety measures will include documentation of adverse events (AE) during and after the procedures.

Follow-ups visits at 3 months and 6 months after the final treatment will be held.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects over 21 years of age seeking treatment and reduction of facial wrinkles
* Subjects should be able understand the investigative nature of the treatment, the possible benefits and side effects, and must sign the Informed Consent Form
* Presence of clearly visible wrinkles in the treated area when the face is relaxed as deemed appropriate by the Investigator
* Subjects willing and able to abstain from partaking in any facial treatments other than the study procedure during study participation
* Willingness to comply with study instructions, to return to the clinic for the required visits, and to have photographs of their face taken

Exclusion Criteria:

* Bacterial or viral infection, acute inflammations
* Impaired immune system
* Isotretinoin in the past 12 months
* Skin related autoimmune diseases
* Radiation therapy and/or chemotherapy
* Poor healing and unhealed wounds in the treatment area
* Metal implants
* Permanent implant in the treated area
* Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body
* Facial dermabrasion, facial resurfacing, or deep chemical peeling in the treatment area within 6 months prior to the treatment
* Current or history of skin cancer, or current condition of any other type of cancer, or pre-malignant moles
* History of any type of cancer
* Active collagen diseases
* Cardiovascular diseases (such as vascular diseases, peripheral arterial disease, thrombophlebitis and thrombosis)
* Pregnancy/nursing or IVF procedure
* History of bleeding coagulopathies, use of anticoagulants
* Any active condition in the treatment area, such as sores, psoriasis, eczema, rash and rosacea
* Any surgical procedure in the treatment area within the last three months or before complete healing
* Poorly controlled endocrine disorders, such as diabetes
* Acute neuralgia and neuropathy
* Kidney or liver failure
* Sensitivity disorders in the treatment area
* Varicose veins, pronounced edemas
* Prior use of dermal fillers, botulinum toxin, lasers, etc. therapies in the treated area that can influence the study results at the investigator discretion
* Unwillingness/inability to not change their usual cosmetics and especially not to use ani-aging or anti-wrinkles products in the treated area during the duration of the study including the follow-up period
* Unwillingness/inability to abstain from cosmetic procedures in the treated area at least 15 days before every examination with the facial image analysis system VISIA
* Any other disease or condition (e.g. eye disease) at the investigator discretion that may pose risk to the patient or compromise the study

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
Assess reduction of wrinkle severity according to the Fitzpatrick Wrinkle and Elastosis Scale | 3 months
  Gathering of clinical evidence that the Device is able to achieve reduction of wrinkle severity according to the Fitzpatrick Wrinkle and Elastosis Scale. The primary efficacy outcome measure is a statistically significant reduction of at least 1.0 score in the average score of Fitzpatrick Wrinkle and Elastosis Scale score according to at least 2 out of 3 blinded dermatologists at 3-months follow-up compared to baseline.

SECONDARY OUTCOMES:
Assess safety profile by recording of adverse events | 7 months
  All AEs including local and systemic reactions not meeting the criteria for "serious adverse events" will be captured on the appropriate CRF. Information to be collected includes event description, time of onset, clinician's assessment of severity, relationship to study product (assessed only by those with the training and authority to make a diagnosis, which would include MD, DDS, DMD, PA, Nurse Practitioner or DO), and time of resolution/stabilization of the event. All AEs occurring during the study must be documented appropriately regardless of relationship to study device. All AEs will be followed to adequate resolution.
Assess subjects' satisfaction with the treatment using Subject Satisfaction Questionnaire | 6 months
  Every subject who completed the treatment will be asked to fill in the Satisfaction Questionnaire at the 3 months follow-up and the 6 months follow-up. This evaluation should reflect overall satisfaction with the results compared to therapy comfort, experienced pain, duration, and application convenience.
  Subjects will be asked: "Overall how are you satisfied with the therapy?" 1 = very satisfied; 2 = satisfied; 3 = neither/nor; 4 = unsatisfied; 5 = very unsatisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Evgeni Hristozov, MD, Principal Investigator — Dermatologist
Locations (1):
- Dermatological center "Lege Artis", Stara Zagora, Bulgaria

IPD SHARING:
Plan to Share IPD: No